CLINICAL TRIAL: NCT05722158
Title: Determination of Bioavailability and Identification of Amino Acid Profile, di- and Tri-peptides in Blood After Oral Ingestion of Collagen Peptides: Randomized, Blinded and Placebo Controlled Clinical Study
Brief Title: Bioavailability of Different Collagen-based Treatments After Oral Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bionos Biotech S.L. (Industry)
Responsible Party: Principal Investigator, José Luis Mullor, Principal Investigator, Bionos Biotech S.L.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Collagen_2022
Record Dates: First submitted 2023-01-18; First posted 2023-02-10 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
Keywords: collagen; bioavailability; peptides; blood; oral; ingestion; randomized; blinded
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): This group will be provided with a placebo solution for comparative purposes.
  Interventions: Dietary Supplement: Dietary supplementation with placebo.
- Collagen-based product CP1 (Experimental): This group will be provided with a the collagen-based product CP1, which will be compared to the placebo group.
  Interventions: Dietary Supplement: Dietary supplementation with the collagen-based product CP1.
- Collagen-based product CP2 (Experimental): This group will be provided with a the collagen-based product CP2, which will be compared to the placebo group.
  Interventions: Dietary Supplement: Dietary supplementation with the collagen-based product CP2.
- Collagen-based product CP3 (Experimental): This group will be provided with a the collagen-based product CP3, which will be compared to the placebo group.
  Interventions: Dietary Supplement: Dietary supplementation with the collagen-based product CP3.
- Collagen-based product CP4 (Experimental): This group will be provided with a the collagen-based product CP4, which will be compared to the placebo group.
  Interventions: Dietary Supplement: Dietary supplementation with the collagen-based product CP4.

INTERVENTIONS:
Dietary Supplement: Dietary supplementation with placebo. — Volunteers will be provided with the placebo. For each volunteer, a blood sample from digital puncture will be obtained, and collagen-derived amino acids, di-peptides and tri-peptides will be quantified by LC-MS.
  Arms: Placebo
Dietary Supplement: Dietary supplementation with the collagen-based product CP1. — Volunteers will be provided with the collagen-derived product CP1. For each volunteer, a blood sample from digital puncture will be obtained, and collagen-derived amino acids, di-peptides and tri-peptides will be quantified by LC-MS.
  Arms: Collagen-based product CP1
Dietary Supplement: Dietary supplementation with the collagen-based product CP2. — Volunteers will be provided with the collagen-derived product CP2. For each volunteer, a blood sample from digital puncture will be obtained, and collagen-derived amino acids, di-peptides and tri-peptides will be quantified by LC-MS.
  Arms: Collagen-based product CP2
Dietary Supplement: Dietary supplementation with the collagen-based product CP3. — Volunteers will be provided with the collagen-derived product CP3. For each volunteer, a blood sample from digital puncture will be obtained, and collagen-derived amino acids, di-peptides and tri-peptides will be quantified by LC-MS.
  Arms: Collagen-based product CP3
Dietary Supplement: Dietary supplementation with the collagen-based product CP4. — Volunteers will be provided with the collagen-derived product CP4. For each volunteer, a blood sample from digital puncture will be obtained, and collagen-derived amino acids, di-peptides and tri-peptides will be quantified by LC-MS.
  Arms: Collagen-based product CP4

SUMMARY:
The goal of this clinical trial is to investigate the postprandial absorption of collagen and elucidate the absorption rate and bioavailability after oral intake of collagen-based products. Participants will be asked to drink solutions containing the study products (one product per group, a total of four products), and blood samples will be obtained by digital puncture at different time points. Plasma will be collected and a set of collagen-derived amino acids, di-peptides and tri-peptides will be quantified by LC-MS. Each product will be compared to the placebo group.

DETAILED DESCRIPTION:
Collagen is characterized by its high content of glycine, proline and hydroxyproline, and it is found to exert beneficial effects on several health benefits. Recent evidence suggests that the consumption of amino acids and/or peptides abundantly present in collagen may have the capacity to influence the synthesis of new collagen in the body. Indeed, it has been found that collagen supplements improve skin moisture, elasticity, and hydration when orally administered. Additionally, collagen reduces the wrinkling and roughness of the skin, and existing studies have not found any side effects of its oral supplements. Thus, to exert any beneficial effects, it is essential that hydrolyzed collagen is optimally absorbed. This study aimed to investigate the postprandial absorption of collagen and elucidate the absorption rate and bioavailability after oral intake.

The study personnel will prepare the drinkable solutions containing the study products in a room accessible to site staff only. Drinkable solutions will be provided to subjects just before consumption. Product ingestion will be early in the morning after overnight fasting for 12 h. On the morning of the experiment, subjects will fast and each subject will take the products orally. Dosage (Quantity of product to consume orally): This is calculated depending on the body weight; 400 mg/kg of body weight with 20 w/v % water. Collagen products (fine powder) will be diluted in water prior consumption. Control group ingest approximately same amount of plain water. Participants cannot drink water within 4 hours before and after the product consumption.

The assessment of the bioavailability of the four collagen-based treatments (CP1, CP2, CP3, CP4) will be evaluated by quantifying 8 di/tri-peptides and the amino acid profile in the blood of 25 volunteers by LC-MS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers to avoid any possible hormonal interference.
* Between 25-45 years old (both included).
* Body weight is 70 kg (60-80 kg (both included), the range depends on the body mass index (BMI). BMI in normal (healthy weight and overweight) range: 18.5 to 29.9 kg/m2. (Reference: WHO and CDC).
* Co-operative and available during the study period.
* Subjects with capacity to understand the purpose and protocol of the study and sign the Informed Consent.

Exclusion Criteria:

* - Diagnosis of allergies to gelatin, red meat (Alpha Gal Syndrome) or fish.
* Diagnosis of diseases about collagen metabolism such as Goodpasture syndrome, scleroderma, periarteritis nodosa or polyarteritis, dermatomyositis, and disseminated lupus erythematosus.
* Diagnosis of following chronic Gastro-Intestinal Tract diseases blocking transfer of polypeptides from GIS to the blood such as: Peptic Ulcer, Duodenal Ulcer, Chronic Atrophic Gastritis, Helicobacter Pylori, Chronic Peptic Disorders, Chronic Acid Reflux = GER and GERD, Celiac Disease, Crohn's Disease, Irritable Bowel Syndrome, Lactose Intolerance, Diverticulitis, Diverticulosis.
* Diagnosis of any diseases such as cardiovascular disease, chronic kidney disease (CKD), gastrointestinal disorder, endocrinological disorder, immunological disorder, metabolic disease.
* Consume more than the recommended alcohol guidelines i.e. >21 alcohol units/week for males and >14 units/week for females (europa.eu).
* Current smoking habit or history of smoking within the past 1 year.
* History of depression, schizophrenia, alcoholism, drug addiction, or mental illness.
* Current or previous intake of contraceptives, female hormones, obesity drugs, absorption inhibitors, antidepressants, or appetite suppressants.
* History of asthma or autoimmune disease Use of oral hormone therapies ie. cortisone or steroids in the 6 months prior to initiation of the study.
* Abnormal liver function or abnormal renal function.
* Blood pressure >140/90 mmHg or hypertension with intake of a diuretic.
* No participation to another clinical trial in the last 6 months.
* No blood donation within a month.
* Problems with overall findings in blood-test results as determined by a specialist.
* Any condition judged by the investigator to be unsuitable for participation in the study.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Quantification of the change of the collagen-derived amino acids, di-peptides and tri-peptides levels in plasma at time 0 minutes (before consuming the product), and 15 minutes, 30 minutes, 120 minutes and 240 minutes after consuming the product. | Upon oral intake, blood samples will be obtained by digital puncture at each time point; Time 0 minutes (before consuming the product), and 15 minutes, 30 minutes, 120 minutes and 240 minutes after consuming the product.
  Upon oral intake, blood samples will be obtained by digital puncture at time 0 minutes (before consuming the product), and 15 minutes, 30 minutes, 120 minutes and 240 minutes after consuming the product. The digital puncture will be performed with Verifine Safety Lancets, and the blood will be collected in MiniCollect tubes. Blood samples will be centrifuged (1000 rpm, 5 minutes, 4ºC) and plasma will be collected. The profile of single amino acids and selected di- and tripeptides will be determined in the plasma samples by mass spectrometry (LC-MS) and the change in the levels of these molecules will be assessed in the specified time points. The following molecules will be analyzed:
  * Single aminoacids (approx. 20 aminoacids, but especially hydroxyproline, glycine, proline)
  * Dipeptides (Pro-Hyp, Hyp-Gly, Ala-Hyp, Phe-Hyp)
  * Tripeptides (Gly-Pro-Hyp, Pro-Hyp-Gly, Ala-Hyp-Gly, Ser-Hyp-Gly)

CONTACTS AND LOCATIONS:
Overall Officials: David Pajuelo Gamez, Principal Investigator — Hospital La Fe
Locations (1):
- Bionos Biotech S.L., Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No